CLINICAL TRIAL: NCT06967168
Title: Feasibility of Developing Personalised Treatment Pathways for Relief of Plantar Heel Pain Using a Sequential Multiple Assignment Randomised Trial (SMART) Study Design
Brief Title: HeEL Pain Pathways Feasibility Study
Acronym: HELPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 8651; RfPPB-22-1937 - Dr Nia Jones (Other Grant/Funding Number: Health and Care Research Wales)
Record Dates: First submitted 2024-01-31; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Plantar Fasciitis
Keywords: pain management; podiatry; musculoskeletal diseases; foot diseases; foot orthoses; extracorporeal shockwave therapy; conservative treatment; self care
MeSH Terms: conditions — Fasciitis, Plantar; Agnosia; Musculoskeletal Diseases; Foot Diseases | interventions — Braces; Foot Orthoses; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomised Trial (SMART)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Adaptive Intervention 1 (outcome subgroups A+B) (Active Comparator): First-line treatment: Virtual consultation. Those whose pain is not resolved after 4 weeks will progress onto second-line treatment: Orthotics.
  Interventions: Behavioral: Virtual consultation; Device: Orthotics
- Adaptive Intervention 2 (outcome subgroups A+C) (Active Comparator): First-line treatment: Virtual consultation. Those whose pain is not resolved after 4 weeks will progress onto second-line treatment: Shockwave therapy (ESWT).
  Interventions: Behavioral: Virtual consultation; Device: Shockwave therapy
- Adaptive Intervention 3 (outcome subgroups D+E) (Active Comparator): First-line treatment: Self-help video. Those whose pain is not resolved after 4 weeks will progress onto second-line treatment: Orthotics.
  Interventions: Behavioral: Self-help video; Device: Orthotics
- Adaptive Intervention 4 (outcome subgroups D+F) (Active Comparator): First-line treatment: Self-help video. Those whose pain is not resolved after 4 weeks will progress onto second-line treatment: Shockwave therapy (ESWT).
  Interventions: Behavioral: Self-help video; Device: Shockwave therapy

INTERVENTIONS:
Behavioral: Virtual consultation — Virtual (telephone) consultation with a podiatrist, who will provide self-management advice to the participant including advice on footwear, massage, and stretching. Supplemented by written advice leaflets.
  Arms: Adaptive Intervention 1 (outcome subgroups A+B); Adaptive Intervention 2 (outcome subgroups A+C)
Behavioral: Self-help video — Self-help video providing self-management advice to the participant including advice on footwear, massage, and stretching. Available online or as a DVD.
  Arms: Adaptive Intervention 3 (outcome subgroups D+E); Adaptive Intervention 4 (outcome subgroups D+F)
Device: Orthotics — Provision of orthotics following an in-person musculoskeletal assessment by a podiatrist to check foot function, footwear, and position of feet, ankles, knees, and hip.
  Podiatrists prescribe, produce, and fit orthotic devices to be worn inside footwear. The devices used in this feasibility study will be selected according to individual patient needs. All will have regulatory certification (CE mark) and will be used in accordance with the manufacturer's Instructions For Use.
  Other Names: Shoe inserts
  Arms: Adaptive Intervention 1 (outcome subgroups A+B); Adaptive Intervention 3 (outcome subgroups D+E)
Device: Shockwave therapy — A 3-week course of Shockwave therapy following an in-person musculoskeletal assessment by a podiatrist to check foot function, footwear, and position of feet, ankles, knees, and hip.
  Extracorporeal shockwave therapy (ESWT) is delivered by a podiatrist in an outpatient clinic. Most patients lie down during the procedure. The machine passes pulses of energy through the skin towards the injured area of the heel. This encourages the body to respond and aims to stimulate the healing process. Participants will need to attend the clinic approximately once a week for three weeks to complete the course of treatment.
  Other Names: ESWT
  Arms: Adaptive Intervention 2 (outcome subgroups A+C); Adaptive Intervention 4 (outcome subgroups D+F)

SUMMARY:
At the moment, no-one is sure what the best way to treat heel pain is. The purpose of this research is to try out some study methods to prepare for a future clinical trial, that will assess how helpful combining different treatments are for people with heel pain (plantar fasciitis). At this stage, the aim is only to test the study processes and ask for feedback - that is why this is called a feasibility study. No experimental techniques or devices will be tested. All of the treatments in the study are routinely carried out in NHS clinics, but participants will be allocated to different combinations of treatments.

Each participant will be asked to complete questionnaires and a diary for around six months in total. Some people will also be invited to take part in an interview or focus group discussion.

DETAILED DESCRIPTION:
This single-centre study will test the feasibility of using a SMART design to provide tailored treatment pathways for people with heel pain. The study will investigate areas of uncertainty relating to the feasibility of a future full-scale SMART study. Key objectives are to assess whether the research design is feasible (including whether enough people can be recruited), and to determine whether the proposed adaptive intervention pathways are acceptable to patients and NHS staff.

50 people with heel pain will be recruited from referrals received by the Podiatry department. Participants will be randomly assigned to two groups initially - half will have a virtual consultation with a podiatrist; the other half will receive a self-help video. After following the advice at home for at least 4 weeks, anyone (in either group) who has not responded to treatment will be offered an assessment in an outpatient clinic. They will then be randomised equally again to receive either an orthotic device (shoe insole) or a course of 'Shockwave therapy' (using a non-invasive device to deliver ultrasound to the injured area).

As well as collecting Patient Reported Outcome Measures (PROMs) for a total duration of 6 months for each participant, process evaluation methods (interviews and focus groups) will be used to talk to patients. They will be asked about their experiences of adaptive intervention pathways and of participating in the feasibility study. The researchers will also interview staff involved in trial design and delivery (clinical members of the study delivery team) about similar topics from a different perspective. Progression criteria will be used to help decide whether to continue with the plan to run a full-scale trial to test effectiveness of the treatment pathways.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or over
* Have symptomatic heel pain (in one or both feet)
* Able to speak, read and understand written and spoken English or Welsh
* Able to provide remote informed consent
* Access to internet and email, or DVD player, with technical support from family, friends or carers if necessary.

Exclusion Criteria:

* Taken part in a prescribed exercise intervention or used prescribed insoles (past 3 months)
* History of major trauma or fracture of the lower leg or below ankle surgery
* Heel pain secondary to a systemic condition/syndrome/malignancy
* Requires ankle-foot orthoses or lower limb device (splint)
* Diabetes or peripheral neuropathy
* History of inflammatory joint disease or autoimmune condition
* Chronic pain syndrome
* Pregnancy
* Pacemaker or other electrical implant
* Blood clotting disorder (haemophilia), blood clot (thrombosis), or current use of anticoagulant medication
* Cortisone injection therapy within the last two weeks
* Unable to complete exercises in self-help resources.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment (Progression Criterion 1) | Through study completion, an average of 1 year.
  Average number of participants per month. Stop if <2; Change if 2-6; Go if >6.
Fidelity of clinical delivery of the correct treatment at the correct stage (Progression Criterion 2) | Through study completion, an average of 1 year.
  Proportion of participants who receive the treatments they are allocated to after each randomisation. Stop if <50%; Change if 50-80%; Go if >80%.
Appropriateness of tailoring criteria and its threshold (Progression Criterion 3) | Through study completion, an average of 1 year.
  Minimum number of participants in any of the SMART outcome subgroups (A-F) at the end of the study. Stop if <1; Change if 1-4; Go if >4.
Rate of retention/loss to follow-up, including withdrawals (Progression Criterion 4) | Through study completion, an average of 1 year.
  Proportion of participants who fail to complete the study. Stop if >50%; Change if 20-50%; Go if <20%.
Acceptability of adaptive intervention pathways amongst patients | Through study completion, an average of 1 year.
  Qualitative interviews and/or focus groups will be carried out with participants to determine the acceptability of adaptive interventions and the study design, including barriers and facilitators to following self-management advice.
Acceptability of adaptive intervention pathways amongst staff | Through study completion, an average of 1 year.
  Qualitative interviews will be carried out with study staff to determine acceptability of adaptive interventions, including barriers and facilitators to delivering the SMART study.

SECONDARY OUTCOMES:
Estimated effect size and variance | Baseline and Week 26
  Composite outcome data from validated PROM - Revised Foot Function Index (short)

OTHER OUTCOMES:
Acceptability of data collection tools (quantitative) | Through study completion, an average of 1 year.
  Completeness of PROM questionnaires and participant diaries/records.
Acceptability of data collection tools (qualitative) | Through study completion, an average of 1 year.
  Qualitative information from staff and participant interviews/focus groups.
Feasibility of collecting health service resource use data (staff time) | Through study completion, an average of 1 year.
  Any deviations from the usual amount of staff time required will be reported in narrative form by the delivery team.
Feasibility of collecting health service resource use data (equipment) | Through study completion, an average of 1 year.
  Any deviations from standard care with respect to the equipment required will be reported in narrative form by the delivery team.
Feasibility of collecting health service resource use data (number of appointments) | Through study completion, an average of 1 year.
  Participants will be invited to indicate their frequency of use of healthcare services in patient diaries. Each week they will be asked how many appointments they have had.
Feasibility of collecting health service resource use data (type of appointment) | Through study completion, an average of 1 year.
  Participants be asked which type(s) of healthcare professional they have had appointments with (GP, nurse, physiotherapist, other) in weekly patient diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Nia J Jones, PhD, Principal Investigator — Cardiff and Vale University Health Board
Locations (1):
- Podiatry Department, Cardiff Royal Infirmary, Cardiff, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No